CLINICAL TRIAL: NCT03789253
Title: Identify Genes/Pathways Responsible for Progression From Low Risk to Higher Risk Prostate Cancer-A New Strategy for Prostate Cancer Prevention
Brief Title: Identify Genes/Pathways Responsible for Progression From Low Risk to Higher Risk Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201712093RINB
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer Stage I
Keywords: active surveillance, microarray, latent, GSEA, latent
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AS cohort with progression: AS cohort with tumor progression
- AS cohort without progression: AS cohort without tumor progression

SUMMARY:
In Taiwan, about 70% of new incident prostate cancer patients have localized disease. Most patients were detected by PSA screening. Among them, many had low-risk PC, which is very likely latent in nature, progresses slowly, and rarely leads to death. Most patients died of other causes, such as other cancers, cardiovascular diseases, and diabetes mellitus. Many guidelines recommend that active surveillance (AS) or watchful waiting (WW) is a good option for low risk patients to avoid overtreatment-related complications. However, 30% of patients on AS will finally need definitive treatments due to disease progression within 10 years. We hypothesize that there are differential gene expressions between progressive and non-progressive tumors. If we can identify key genes or pathways that are responsible for progression of low risk PC to higher risk diseases, PC progression could be reduced substantially by regulating these genes or pathways and maintain long-term cancer latency to control non-metastatic PC. In light of the high prevalence rate of latent PC in adult men, the strategy is in fact the best strategy for preventing clinical PC.

DETAILED DESCRIPTION:
At the Department of Urology, NTUH, we have established a largest Chinese AS/WW cohort, which were prospectively collected since 2013. There were already 280 AS and 100 WW patients. Most AS patients have undergone serial prostate re-biopsies every 1 to 2 years, which is actually our cutting edge in the field. 87 men had at least twice biopsies at our hospital (mean interval 15 months). 26 of them showed pathological progression (Group As) who have been treated aggressively. The other 61 men had no progression even after multiple biopsies (Group Bs). So, we may compare the genetic changes in each subject in Group A to reveal genetic changes responsible for progression. We can also compare baseline expressions between Group A and B to predict progression. We also can correlate genetic alterations in Group A with cancer phenotypes and short-term post-treatment outcomes.

Here are the four Specific Aims:

Aim-1. To investigate the role of known genes or pathways in mediating progression from low risk to higher risk by using serial biopsy paraffin embedded tissue blocks from our AS patients. These known genes/pathways are selected from published reports, which are found to be related to progression from low to higher grade PC, such as Ki-67, PTEN loss, and chromosome 8 alterations.

Aim-2. There was only one cDNA microarray gene bank (GSE37199) published in the literature (Lancet Oncol. 2012; 13:1114) that was associated with differential expression between AS and mCRPC cohorts. We will proceed with the Gene Set Enrichment Analysis (GSEA) to identify more potential genes or pathways that have NOT been specifically demonstrated relating to AS progression. These new genes or pathways will then be studied in Aim-1.

Aim-3. We will perform global cDNA microarray sing non-cancer part of the serial biopsy paraffin tissue blocks from our AS cohort, followed by GSEA to reveal differential gene expression between Group A and B patients. Hopefully we can identify genes/pathways that are related to progression of low risk or latent PC in Taiwanese.

Aim-4. To conduct multivariate analyses considering not only key genetic alterations but also multiple clinicopathological parameters to build up a model predicting progression from low to higher risk PC.

In fact, the only one published study (Lancet Oncol. 2012;13:1114) was to reveal differential cDNA expression in blood cells between AS and mCRPC cohorts, but not between progressive and non-progressive patients. Therefore, the study design was defective because the obtained differential expression may not reflect what really happened in low risk cancer progression. To our knowledge, there has been no differential genetic expression study or the GSEA study for AS cohort. In addition, we have the largest Taiwanese/Chinese cohort on AS/WW and abundant serial biopsy specimens. In summary, our study which focuses on genomic research on AS cohort is a new strategy to prevent clinical PC and is of high novelty and clinical implications.

ELIGIBILITY:
Inclusion Criteria:

1. Historically or cytologically confirmed adenocarcinoma of prostate.
2. Have or ever received active Surveillance as the main conservative management at NTUH (National Taiwan University Hospital).
3. Have or will receive prostate biopsy to confirm tumor progression after the diagnosis of prostate cancer.

Exclusion Criteria:

1. Have received systemic chemotherapy, pelvic radiotherapy or androgen deprivation therapy (ADT) before the obtainment of pathological specimen from prostate operation or biopsy.
2. Subjects who disagree with signing the informed consent.

Ages: 40 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low or intermediate risk prostate cancer patients receiving active surveillance
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Gene expression | 3 years
  Using GESA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No